CLINICAL TRIAL: NCT02868086
Title: The Impact of Two Strategies in the Monitoring of Exudative ARMD on the Visual Acuity (by OCT B Scan or OCT Angiography)
Acronym: REPERM-OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMT_2015_42
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related macular degeneration; Optical coherence tomography angiography
MeSH Terms: conditions — Macular Degeneration

ARMS (2):
- Tested patients (Experimental): Patients treated with anti-angiogenics for ARMD : monitoring using optical coherence tomography angiography
  Interventions: Device: OCT angiography
- Control patients (Active Comparator): Patients treated with anti-angiogenics for ARMD : monitoring during common practice via optical coherence tomography B scans
  Interventions: Device: OCT B-scans

INTERVENTIONS:
Device: OCT B-scans
  Arms: Control patients
Device: OCT angiography
  Arms: Tested patients

SUMMARY:
The treatment of neovascular age-related macular degeneration (ARMD) is a major issue of public health. The therapeutic arsenal has widely grown throughout the years with the emergence of intra-vitreous anti-angiogenic treatments, under different surveillance protocols. The "PRN" surveillance (pro re nata: an on-demand treatment with monthly follow-up) allows a faster re-injection in case of neovascular relapse in order to maintain the best visual acuity. This therapeutic protocol is guided by the sub-retinal neovascular signs of activity. The monitoring is done during common practice via OCT B scans showing indirect signs of neovascular activity (exudation signs). OCT retinal imaging has been recently enriched with new programs allowing the visualization of sub-retinal neovessels without the use dyes (OCT angiography). The OCT angiography is automatically done by a program using standard OCT sections. During the monitoring of a patient using the OCT A, the signs of renewed neovascular activity are represented by an "arterialization" or the development of an arteriole network of the neovessel with the reappearance of a hyper reflective flow after a neovascular regressive phase. Indeed, the visualization of neovessels during the monitoring by Angio-OCT may lead to therapeutical modifications (anticipation of the injections). Knowing that the injection time-table of ARMD patients treated with anti-angiogenics is determined by sub-retinal neovascular signs of activity. This activity is evaluated during routine clinical practice by very specific signs, observable on OCT B scans. The hypothesis of this study is that the search of activity sins on the Angio-OCT, a new technic of image analysis performed on the OCT, may modify this injection time-table, with an impact of the patient's visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 50 years old
* with exudative ARMD,
* treated with intra-vitreous anti-angiogenics following a PRN protocol (pro re nata)
* Absence of atrophy of the central pigment epithelium

Exclusion Criteria

* Opposition to participate in this research
* Persons enjoying legal protection measure
* Lack of affiliation to social security and universal health coverage
* Pregnant or lactating
* Another cause of Choroidal neovascularization
* Unbalanced glaucoma
* Eye surgery less than 3 months on the studied eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement or stabilization | Between the inclusion and 1 year of follow-up
  Proportion of patients with visual acuity improvement or stabilization

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France

REFERENCES:
- [Result] Sukkarieh G, Vasseur V, Lejoyeux R, Wolff B, Mauget-Faysse M. One-year outcome of neovascular age-related macular degeneration patients followed-up using different optical coherence tomography modalities. Eur J Ophthalmol. 2022 Nov;32(6):3503-3509. doi: 10.1177/11206721221088260. Epub 2022 Mar 14. PMID 35285308